CLINICAL TRIAL: NCT04710992
Title: Influence of Percutaneous Electrolysis on Endogenous Pain Modulation: A Randomized Clinical Trial
Brief Title: Influence of Percutaneous Electrolysis on Endogenous Pain Modulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Sergio Varela Rodríguez, PhD candidate, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Electrolysis550
Record Dates: First submitted 2021-01-10; First posted 2021-01-15 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Pain
Keywords: Electric Stimulation Therapy; Randomized Clinical Trial; Interventional Ultrasonography; Percutaneous Electrolysis; Endogenous Pain Modulation; Pain; Conditioned Pain Modulation; Sensory Thresholds
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Needling Group (Sham Comparator): The needle will be inserted for 90 seconds without galvanic current.
  Interventions: Procedure: Isolated needling procedure
- Low intensity percutaneous electrolysis (Experimental): A single impact of galvanic current will be applied with an intensity of 0.3 mA for 90 seconds.
  Interventions: Procedure: Low intensity percutaneous electrolysis
- High intensity percutaneous electrolysis (Experimental): Three impacts of galvanic current will be applied with an intensity of 3 mA and a duration of 3 seconds each.
  Interventions: Procedure: High intensity percutaneous electrolysis

INTERVENTIONS:
Procedure: Isolated needling procedure — The needle will be inserted into the common extensor tendon of the epicondyle (dominant elbow) for 90 seconds without galvanic current.
  Arms: Needling Group
Procedure: Low intensity percutaneous electrolysis — Once the needle is located in the common extensor tendon of the epicondyle (dominant elbow), a single impact of galvanic current will be applied with an intensity of 0.3 mA for 90 seconds.
  Arms: Low intensity percutaneous electrolysis
Procedure: High intensity percutaneous electrolysis — The needle will be inserted in the target position during the same time as in the other groups (90 seconds). During the first stage of intervention the needle will be imbedded without galvanic current and when the end of the application time approaches (approximately 75 seconds) three impacts of galvanic current will be applied with an intensity of 3 mA and a duration of 3 seconds each.
  Arms: High intensity percutaneous electrolysis

SUMMARY:
Percutaneous electrolysis is a minimally invasive approach that consists in the application of a galvanic current through an acupuncture needle. Although several mechanisms and effects are attributed to percutaneous electrolysis, currently there are only a few publications that delve into this topic. The aim of this study is to investigate the influence of percutaneous electrolysis on the endogenous pain modulation. Four groups of intervention will be involved: no-intervention, isolated needling procedure, low intensity percutaneous electrolysis and high intensity percutaneous electrolysis. The effects on the pain modulation system will be evaluated before and immediately after the intervention, through pressure pain thresholds, conditioned pain modulation and temporal summation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy asymptomatic subjects
* Aged 18 to 40 years
* Both genders

Exclusion Criteria:

* Belonephobia or fear of needles
* Neurological, cardiovascular or metabolic diseases
* Any pathology or process that causes pain
* Cutaneous alterations
* Pregnancy
* Cognitive and sensitivity disorders
* Fibromyalgia
* Frequent or recent (24 hours before) intake of alcohol and other drugs
* Have received pharmacological, physiotherapeutic or other treatment in the last week
* Intake of caffeine in the two hours prior to measurement
* Vigorous physical activity on the day of testing

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline Conditioned Pain Modulation (evaluated by pressure algometry) immediately after the intervention | Baseline and immediately after the intervention
  Assessed by algometry. Conditioning stimulus: pressure cuff on the arm. Measured at three locations (bilaterally): common extensor tendon of the epicondyle, cervical spine and tibialis anterior muscle.

SECONDARY OUTCOMES:
Change from baseline Pressure Pain Thresholds immediately after the intervention | Baseline and immediately after the intervention
  Assessed by algometry. Measured at three locations (bilaterally): common extensor tendon of the epicondyle, cervical spine and tibialis anterior muscle.
Change from baseline Temporal Summation (evaluated by VNRS) immediately after the intervention | Baseline and immediately after the intervention
  Assessed by Verbal Numeric Rating Scale (11-point). Temporary stimuli: 10 consecutive pressures with the algometer at the intensity of the pressure pain threshold. Three locations (bilaterally): common extensor tendon of the epicondyle, cervical spine and tibialis anterior muscle.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Enfermería y Fisioterapia de la Universidad de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garcia Bermejo P, De La Cruz Torres B, Naranjo Orellana J, Albornoz Cabello M. Autonomic Responses to Ultrasound-Guided Percutaneous Needle Electrolysis: Effect of Needle Puncture or Electrical Current? J Altern Complement Med. 2018 Jan;24(1):69-75. doi: 10.1089/acm.2016.0339. Epub 2017 Jan 30. PMID 28135129
- [Background] Valera-Garrido F, Minaya-Munoz F, Medina-Mirapeix F. Ultrasound-guided percutaneous needle electrolysis in chronic lateral epicondylitis: short-term and long-term results. Acupunct Med. 2014 Dec;32(6):446-54. doi: 10.1136/acupmed-2014-010619. Epub 2014 Aug 13. PMID 25122629
- [Background] Abat F, Diesel WJ, Gelber PE, Polidori F, Monllau JC, Sanchez-Ibanez JM. Effectiveness of the Intratissue Percutaneous Electrolysis (EPI(R)) technique and isoinertial eccentric exercise in the treatment of patellar tendinopathy at two years follow-up. Muscles Ligaments Tendons J. 2014 Jul 14;4(2):188-93. eCollection 2014 Apr. PMID 25332934
- [Background] Nir RR, Yarnitsky D. Conditioned pain modulation. Curr Opin Support Palliat Care. 2015 Jun;9(2):131-7. doi: 10.1097/SPC.0000000000000126. PMID 25699686
- [Background] Fernandez-de-Las-Penas C, Nijs J. Trigger point dry needling for the treatment of myofascial pain syndrome: current perspectives within a pain neuroscience paradigm. J Pain Res. 2019 Jun 18;12:1899-1911. doi: 10.2147/JPR.S154728. eCollection 2019. PMID 31354339
- [Background] Damien J, Colloca L, Bellei-Rodriguez CE, Marchand S. Pain Modulation: From Conditioned Pain Modulation to Placebo and Nocebo Effects in Experimental and Clinical Pain. Int Rev Neurobiol. 2018;139:255-296. doi: 10.1016/bs.irn.2018.07.024. Epub 2018 Aug 14. PMID 30146050
- [Derived] Sanchez-Gonzalez JL, Navarro-Lopez V, Calderon-Diez L, Varela-Rodriguez S, Fernandez-de-Las-Penas C, Sanchez-Sanchez JL. Effectiveness of different percutaneous electrolysis protocols in the endogenous modulation of pain: A Double-Blinded Randomized Clinical Trial. Musculoskelet Sci Pract. 2023 Nov;68:102872. doi: 10.1016/j.msksp.2023.102872. Epub 2023 Oct 11. PMID 37847947